CLINICAL TRIAL: NCT04394962
Title: The Use of Virtual Reality Technology in Infertile Women Undergoing in Vitro Fertilization-embryo Transfer: A Randomized Controlled Trial
Brief Title: Virtual Reality Use in Assisted Reproductive Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr cliff Librach (Other)
Responsible Party: Sponsor-Investigator, Dr cliff Librach, Clifford Librach, MD, FRCS(C), FACOG(REI), Director of the Create Fertility Centre, Professor, Department of Obstetrics and Gynecology, University of Toronto, Create Fertility Center
Organization: Create Fertility Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CL1E
Record Dates: First submitted 2020-05-06; First posted 2020-05-20 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: IVF Outcomes; Stress Levels
Keywords: Virtual reality; In vitro fertilization; Embryo transfer

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The Physician performing the embryo transfer will be blinded to the patient's group randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients who will be randomized to the control group will be waiting for the ET procedure without any intervention and without any deviation from the standard of care
- Study group (Experimental): Exposure to virtual reality environment exposure
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Patients randomized to the study group, will be provided with the VR headset and sensors. The VR exposure will take place before the ET procedure, during their routine pre-transfer waiting period, in a private room. The patient will be able to choose between three different calming VR environments (3 scenes: beach sunset, palm tree patio or redwood forest) and will be exposed to the chosen VR environment for a continuous duration of 15-30 minutes. The VR exposure will be passive, and the patient can control her observation inside the environment by herself, simply by moving her head. During this period, at any time and for any reason, the patient can discontinue the use of the VR session simply by self-removing the helmet
  Other Names: "Oculus Rift" system; Immersive environment
  Arms: Study group

SUMMARY:
The study will examine the effect of exposure to virtual reality on stress levels and pregnancy rates, in infertile women undergoing in vitro fertilization embryo transfer

DETAILED DESCRIPTION:
In vitro fertilization (IVF) treatment involving ovarian stimulation, oocyte retrieval and embryo transfer (ET) is an effective treatment for various causes of infertility. Despite advances in ovarian stimulation regimens and laboratory conditions, many IVF cycles do not result in pregnancy, and repeated treatment cycles are required. According to the latest Assisted reproductive technology (ART) surveillance report in the United states, of 143,286 procedures that progressed to the ET stage, 50.9% resulted in a pregnancy and 41.4% in a live-birth. Achieving higher pregnancy and live birth rates remains a leading priority of IVF units worldwide. Both IVF practitioners and patients keep searching for new ways to improve reproductive outcomes.

IVF is a multidimensional stressor. The treatment itself constitutes the primary stressor and is most likely to evoke anxiety. The highest anxiety scores were experienced before embryo transfer and were comparable to anxiety scores obtained from surgical female patients in the immediate preoperative period. Hence, it is not surprising that ET is defined by many investigators as a crucial event for determining IVF outcome, and many patients perceive it as the culmination of the IVF treatment. The stress this procedure may cause can result in a variety of autonomous nervous system expressions, altered uterine gene expression, resulting in decreased uterine receptivity, or an increase in uterine contraction frequency, which may be inversely correlated to embryo implantation and pregnancy rates in IVF. Several studies found that women who did not become pregnant with IVF, reported experiencing more stress during treatment than those who achieved pregnancy.

Although the exact mechanism whereby stress interferes with reproductive processes is not fully understood, experimental evidence increasingly indicates that lower stress levels result in better fertility treatment outcome.

The use of complementary medicine or adjuvant therapies to reduce psychological stress during ART therapy and improve IVF outcomes is increasing. Various alternative therapies have been proposed to improve reproductive outcomes during IVF treatment, such as acupuncture and Chinese herbal medicines. However, the impact of these therapies on IVF outcomes was inconclusive.

The impact of medical clowning as a stress-reducing technique for 12-15 minutes after ET was found to increase the pregnancy rate - 36.4% in the intervention group compared with 20.2% in the control group. Other interventions, specifically prior or during the IVF-ET procedure itself have been studied in the context of improving cycle outcome and/or reducing anxiety levels.

In order to assess anxiety levels before and after interventions, most of these studies included the validated "State-Trait Anxiety Inventory" (STAI) questionnaire, which is a self-assessment questionnaire, consisting of 40 items rated on 4-point Likert scale. The scale consists of two sub-dimensions: the "state anxiety" has 20 items and is used to determine what is felt at a specific moment under certain conditions, and the "trait anxiety" has 20 items and is used to determine what has been felt in the last seven days. Higher scores are positively correlated with higher levels of anxiety. Other studies assessing stress related to ET procedure used salivary a-amylase (SAA). SAA measurement presents a non-invasive and a highly reliable indicator of sympathetic-adrenal medullary activity can be used as a physiologic indicator of the acute stress response.

The impact of hypnosis during ET on the outcome of IVF was studied in 89 patients, compared with controls. The results suggested that the use of hypnosis during ET may significantly improve the IVF-ET cycle outcome in terms of increased implantation rates (IR) and clinical pregnancy rates (CPR).

Harp therapy during ET of 90 IVF patients was found to significantly decrease levels of anxiety post transfer and having a positive effect on acute levels of stress, compared with controls. However, CPR was comparable between the harp group and the control group. Another study assessed the effectiveness of a deep relaxation massage therapy prior to frozen ET in 56 IVF patients. In patients using the massage therapy prior to ET, statistically significant increases in pregnancy and live birth rates were observed when compared with the control group (58.9% vs 41.7%, and 32.0% vs 20.3%, respectively). The researchers hypothesized these improvements were most likely due to a relaxing effect on patients and reduction in stress, leading to a reduction in uterine contractions.

A recent randomized controlled trial assessed the effect of music therapy in women undergoing IVF-ET. They examined the effect of music therapy before and after ET, on the anxiety levels and pregnancy rates in 89 IVF patients. The mean state anxiety scores decreased in both groups, however these changes did not reach statistical significance. CPR were comparable between the groups.

Virtual reality (VR) is a therapeutic approach which has been gaining attention over the past two decades for both medical and psychiatric purposes. VR is an advanced technological system that allows users to be transported into a 'virtual world'. Users are engaged in a fully immersive VR experience through a combination of technologies, including a head-mounted display, headphones with sound/music and noise reduction, and another device for manipulation/navigation of the virtual environment. Multimodal stimuli contribute to a sense of actual presence/immersion in the virtual world, thus making the VR experience distinct from a passive visual or auditory stimuli. Being a safe, non-invasive and easy to use technique, VR therapy has been explored for numerous health applications, showing positive outcomes in clinical conditions such as anxiety disorders, addictions, phobias, posttraumatic stress disorder, eating disorders, stroke rehabilitation, and pain management. A recent systematic review including 11 VR studies and 467 patients, concluded that VR's immersive, entertaining effects are useful for redirecting the patient's attention away from painful treatment experiences and reducing anxiety, discomfort, or unpleasantness. Other studies also showed a significant decrease in pain perception and state anxiety scores when treated with VR, as indicated by anxiety questionnaires, pulse rate reduction, and electroencephalogram (EEG) changes when treated with VR as compared with controls, all supporting the therapeutic potential of VR for anxiety management and stress reduction.

A study presented at the 2018 anesthesia congress in Europe (Unpublished data) compared the effect of two different VR sessions (distraction and hypnosis) before sedation, on the anxiety level and the following cycle outcomes in 100 IVF patients. The preliminary results of the study showed a reduction in the anxiety scores in both groups, however the differences between the groups did not reach statistical significance.

The aim of this study is to examine the effects of VR technology on the most stressful event during IVF-the transfer of embryos into the uterus. The investigators will use the STAI questionnaire to assess levels of anxiety experienced during the ET procedure, in participants exposed to VR session before the ET, compared with participants who are not exposed.

The investigators hypothesize that the use of this unique technology before the procedure may reduce stress levels and consequently improve implantation and pregnancy rates.

According to a recent literature review, there are no published studies examining the effect of VR prior to ET on IVF outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 21-45-year-old female patients, if using own ovum. Patients above this age range may be approached for study if using a donated ovum, as long as "egg age" (age of donor at ovum pick up) falls in 21-45 age range.
* Undergoing frozen ET procedures, and approached for study on "Day 2 - Day 4" of ET transfer cycle.
* Ability to provide written consent to use VR technology before the ET procedure

Exclusion Criteria:

* Contraindication to use VR technology (Epilepsy/previous seizure, claustrophobia, current migraine, heart disease, visual and/or auditory deficits/use of medical devices such as cardiac pacemaker or hearing aids)
* Anxiety disorder and/or Regular use of anti-anxiety medications
* Major uterine anomalies and/or uterine fibroids distorting the cavity

Ages: 21 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate (CPR) | Assessed 4 weeks after ET (= 6 weeks of gestation)
  The difference in CPR (determined by sonographic evidence of a gestational sac and fetal heart rate at 6 weeks' gestation by transvaginal ultrasound) between the study and the control group. An increase of 15% in the clinical pregnancy rate in the study group will be considered as significant.

SECONDARY OUTCOMES:
Stress levels - STAI questionnaires | Questionnaires will be filled out in 3 different time points during the study: 1) Day 1 of recruitment, before beginning the medications for endometrial preparation 2) ET day, 30-60 minutes before ET 3) ET day, 5-10 minutes after ET procedure
  Will be assessed using the STAI questionnaire (scored 20-80 points). We are expecting a 25% decrease in the STAI scores in the study group to be significant, based on clinical experience with similar patient population
Salivary alpha amylase (SAA) levels | Samples will be collected in 3 different time points during the study: 1) Day 1 of recruitment, before beginning the medications for endometrial preparation 2) ET day, 30-60 minutes before ET 3) ET day, 5-10 minutes after ET procedure
  Salivary samples will be collected and analyzed. A 30% decrease in the SAA levels in the study group vs control will be considered significant, based on a previous study
Sympathetic autonomous nervous system expressions | Measurements will be taken in 3 different time points during the study: 1) Day 1 of recruitment, before beginning the medications for endometrial preparation 2) 30-60 minutes before ET 3) ET day, 5-10 minutes after ET procedure
  Heart rate & blood pressure measurements. These 2 sympathetic nervous system variables were selected as physical parameters which may indicate anxiety. A significant change between the groups will be based on clinical experience with similar patient populations. An estimated one-third (33%) of the patients would experience elevated blood pressure and/or heart rate readings in the moderate-to-severe range during the standard procedure. VR exposure therapy is expected to reduce this proportion to 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Librach, MD, Principal Investigator — CReATe Fertility Centre
Locations (1):
- Create Fertility Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sunderam S, Kissin DM, Crawford SB, Folger SG, Boulet SL, Warner L, Barfield WD. Assisted Reproductive Technology Surveillance - United States, 2015. MMWR Surveill Summ. 2018 Feb 16;67(3):1-28. doi: 10.15585/mmwr.ss6703a1. PMID 29447147
- [Background] Porat-Katz A, Eldar-Geva T, Kahane A, Laufer N, Younis JS, Radin O, Paltiel O. Use of complementary medical therapies by Israeli patients undergoing in vitro fertilization. Int J Gynaecol Obstet. 2015 May;129(2):133-7. doi: 10.1016/j.ijgo.2014.11.021. Epub 2015 Feb 7. PMID 25687239
- [Background] Verhaak CM, Smeenk JM, Evers AW, Kremer JA, Kraaimaat FW, Braat DD. Women's emotional adjustment to IVF: a systematic review of 25 years of research. Hum Reprod Update. 2007 Jan-Feb;13(1):27-36. doi: 10.1093/humupd/dml040. Epub 2006 Aug 29. PMID 16940360
- [Background] Yong P, Martin C, Thong J. A comparison of psychological functioning in women at different stages of in vitro fertilization treatment using the mean affect adjective check list. J Assist Reprod Genet. 2000 Nov;17(10):553-6. doi: 10.1023/a:1026429712794. PMID 11209535
- [Background] Kondoh E, Okamoto T, Higuchi T, Tatsumi K, Baba T, Murphy SK, Takakura K, Konishi I, Fujii S. Stress affects uterine receptivity through an ovarian-independent pathway. Hum Reprod. 2009 Apr;24(4):945-53. doi: 10.1093/humrep/den461. Epub 2008 Dec 20. PMID 19098291
- [Background] Levitas E, Parmet A, Lunenfeld E, Bentov Y, Burstein E, Friger M, Potashnik G. Impact of hypnosis during embryo transfer on the outcome of in vitro fertilization-embryo transfer: a case-control study. Fertil Steril. 2006 May;85(5):1404-8. doi: 10.1016/j.fertnstert.2005.10.035. Epub 2006 Mar 29. PMID 16566936
- [Background] Fanchin R, Righini C, de Ziegler D, Olivennes F, Ledee N, Frydman R. Effects of vaginal progesterone administration on uterine contractility at the time of embryo transfer. Fertil Steril. 2001 Jun;75(6):1136-40. doi: 10.1016/s0015-0282(01)01787-3. PMID 11384639
- [Background] Fanchin R, Righini C, Olivennes F, Taylor S, de Ziegler D, Frydman R. Uterine contractions at the time of embryo transfer alter pregnancy rates after in-vitro fertilization. Hum Reprod. 1998 Jul;13(7):1968-74. doi: 10.1093/humrep/13.7.1968. PMID 9740459
- [Background] Zhu L, Che HS, Xiao L, Li YP. Uterine peristalsis before embryo transfer affects the chance of clinical pregnancy in fresh and frozen-thawed embryo transfer cycles. Hum Reprod. 2014 Jun;29(6):1238-43. doi: 10.1093/humrep/deu058. Epub 2014 Mar 23. PMID 24664129
- [Background] Boivin J, Takefman JE. Stress level across stages of in vitro fertilization in subsequently pregnant and nonpregnant women. Fertil Steril. 1995 Oct;64(4):802-10. doi: 10.1016/s0015-0282(16)57858-3. PMID 7672154
- [Background] Csemiczky G, Landgren BM, Collins A. The influence of stress and state anxiety on the outcome of IVF-treatment: psychological and endocrinological assessment of Swedish women entering IVF-treatment. Acta Obstet Gynecol Scand. 2000 Feb;79(2):113-8. doi: 10.1034/j.1600-0412.2000.079002113.x. PMID 10696958
- [Background] Eugster A, Vingerhoets AJ, van Heck GL, Merkus JM. The effect of episodic anxiety on an in vitro fertilization and intracytoplasmic sperm injection treatment outcome: a pilot study. J Psychosom Obstet Gynaecol. 2004 Mar;25(1):57-65. doi: 10.1080/01674820410001737441. PMID 15376405
- [Background] Friedler S, Glasser S, Azani L, Freedman LS, Raziel A, Strassburger D, Ron-El R, Lerner-Geva L. The effect of medical clowning on pregnancy rates after in vitro fertilization and embryo transfer. Fertil Steril. 2011 May;95(6):2127-30. doi: 10.1016/j.fertnstert.2010.12.016. Epub 2011 Jan 6. PMID 21211796
- [Background] Manheimer E, van der Windt D, Cheng K, Stafford K, Liu J, Tierney J, Lao L, Berman BM, Langenberg P, Bouter LM. The effects of acupuncture on rates of clinical pregnancy among women undergoing in vitro fertilization: a systematic review and meta-analysis. Hum Reprod Update. 2013 Nov-Dec;19(6):696-713. doi: 10.1093/humupd/dmt026. Epub 2013 Jun 27. PMID 23814102
- [Background] Qian Y, Xia XR, Ochin H, Huang C, Gao C, Gao L, Cui YG, Liu JY, Meng Y. Therapeutic effect of acupuncture on the outcomes of in vitro fertilization: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 Mar;295(3):543-558. doi: 10.1007/s00404-016-4255-y. Epub 2016 Dec 19. PMID 27995371
- [Background] Wang X, Lin H, Chen M, Wang J, Jin Y. Effect of acupuncture on in vitro fertilization: An updated systematic review and data mining protocol. Medicine (Baltimore). 2018 Jun;97(24):e10998. doi: 10.1097/MD.0000000000010998. PMID 29901590
- [Background] Villahermosa DI, Santos LG, Nogueira MB, Vilarino FL, Barbosa CP. Influence of acupuncture on the outcomes of in vitro fertilisation when embryo implantation has failed: a prospective randomised controlled clinical trial. Acupunct Med. 2013 Jun;31(2):157-61. doi: 10.1136/acupmed-2012-010269. Epub 2013 Mar 19. PMID 23512550
- [Background] Spielberger CD. Manual for the State-Trait Anxiety Inventory: STAI (form Y). Palo Alto, CA: Consulting Psychologists Press. 1983.
- [Background] Murphy EM, Nichols J, Somkuti SG, Sobel M, Braverman A, Barmat LI. Randomized trial of harp therapy during in vitro fertilization-embryo transfer. J Evid Based Complementary Altern Med. 2014 Apr;19(2):93-8. doi: 10.1177/2156587213514054. Epub 2013 Dec 18. PMID 24668261
- [Background] Cheung C, Saravelos SH, Chan T, Sahota DS, Wang CC, Chung PW, Li TC. A prospective observational study on the stress levels at the time of embryo transfer and pregnancy testing following in vitro fertilisation treatment: a comparison between women with different treatment outcomes. BJOG. 2019 Jan;126(2):271-279. doi: 10.1111/1471-0528.15434. Epub 2018 Sep 25. PMID 30106234
- [Background] Saravelos SH, Wong AW, Kong GW, Huang J, Klitzman R, Li TC. Pain during embryo transfer is independently associated with clinical pregnancy in fresh/frozen assisted reproductive technology cycles. J Obstet Gynaecol Res. 2016 Jun;42(6):684-93. doi: 10.1111/jog.12962. Epub 2016 Feb 24. PMID 26916559
- [Background] McKay KA, Buen JE, Bohan KJ, Maye JP. Determining the relationship of acute stress, anxiety, and salivary alpha-amylase level with performance of student nurse anesthetists during human-based anesthesia simulator training. AANA J. 2010 Aug;78(4):301-9. PMID 20879631
- [Background] Aba YA, Avci D, Guzel Y, Ozcelik SK, Gurtekin B. Effect of music therapy on the anxiety levels and pregnancy rate of women undergoing in vitro fertilization-embryo transfer: A randomized controlled trial. Appl Nurs Res. 2017 Aug;36:19-24. doi: 10.1016/j.apnr.2017.05.005. Epub 2017 May 22. PMID 28720234
- [Background] Okhowat J, Murtinger M, Schuff M, Wogatzky J, Spitzer D, Vanderzwalmen P, Wirleitner B, Zech NH. Massage therapy improves in vitro fertilization outcome in patients undergoing blastocyst transfer in a cryo-cycle. Altern Ther Health Med. 2015 Mar-Apr;21(2):16-22. PMID 25830275
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Background] Niharika P, Reddy NV, Srujana P, Srikanth K, Daneswari V, Geetha KS. Effects of distraction using virtual reality technology on pain perception and anxiety levels in children during pulp therapy of primary molars. J Indian Soc Pedod Prev Dent. 2018 Oct-Dec;36(4):364-369. doi: 10.4103/JISPPD.JISPPD_1158_17. PMID 30324926
- [Background] Garrett B, Taverner T, Gromala D, Tao G, Cordingley E, Sun C. Virtual Reality Clinical Research: Promises and Challenges. JMIR Serious Games. 2018 Oct 17;6(4):e10839. doi: 10.2196/10839. PMID 30333096
- [Background] Dascal J, Reid M, IsHak WW, Spiegel B, Recacho J, Rosen B, Danovitch I. Virtual Reality and Medical Inpatients: A Systematic Review of Randomized, Controlled Trials. Innov Clin Neurosci. 2017 Feb 1;14(1-2):14-21. eCollection 2017 Jan-Feb. PMID 28386517
- [Background] Gershon J, Zimand E, Lemos R, Rothbaum BO, Hodges L. Use of virtual reality as a distractor for painful procedures in a patient with pediatric cancer: a case study. Cyberpsychol Behav. 2003 Dec;6(6):657-61. doi: 10.1089/109493103322725450. PMID 14756933
- [Background] Tarrant J, Viczko J, Cope H. Virtual Reality for Anxiety Reduction Demonstrated by Quantitative EEG: A Pilot Study. Front Psychol. 2018 Jul 24;9:1280. doi: 10.3389/fpsyg.2018.01280. eCollection 2018. PMID 30087642
- [Background] Patterson DR, Tininenko JR, Schmidt AE, Sharar SR. Virtual reality hypnosis: a case report. Int J Clin Exp Hypn. 2004 Jan;52(1):27-38. doi: 10.1076/iceh.52.1.27.23925. PMID 14768967